CLINICAL TRIAL: NCT02008916
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study of Secukinumab to Demonstrate the Efficacy at 16 Weeks and to Assess the Long-term Safety, Tolerability and Efficacy up to 3 Years in Subjects With Active Ankylosing Spondylitis
Brief Title: 16-week Efficacy and 3-year Safety, Tolerability and Efficacy of Secukinumab in Active Ankylosing Spondylitis Patients
Acronym: MEASURE 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2314; 2013-001090-24 (EudraCT Number)
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Spondylitis, Ankylosing
Keywords: AIN457, ankylosing spondylitis, chronic inflammatory disease, inflammatory back pain, secukinumab, self-injection
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Secukinumab 10 mg/kg i.v. / 300 mg s.c. (Experimental): Three i.v. infusions: at Baseline and weeks 2 and 4, followed by one s.c. injection every four weeks until the end of the study.
  Interventions: Drug: Secukinumab
- Secukinumab 10 mg/kg i.v. / 150 mg s.c. (Experimental): Three i.v. infusions: at Baseline and weeks 2 and 4, followed by one s.c. injection every four weeks until the end of the study.
  Interventions: Drug: Secukinumab
- Placebo i.v. and s.c. (Placebo Comparator): Three i.v. infusions: at Baseline and weeks 2 and 4, followed by one s.c. injection at weeks 8 and 12. At week 16, patients were re-randomised to one of the active treatment arms, to receive secukinumab s.c. Q4W until the end of the study.
  Interventions: Drug: Placebo secukinumab

INTERVENTIONS:
Drug: Secukinumab — AIN457 (Secukinumab) is a human monoclonal antibody. Secukinumab binds and reduces the activity of Interleukin 17 (IL-17).
  Other Names: AIN457
  Arms: Secukinumab 10 mg/kg i.v. / 150 mg s.c.; Secukinumab 10 mg/kg i.v. / 300 mg s.c.
Drug: Placebo secukinumab — Placebo to AIN457 (Secukinumab)
  Arms: Placebo i.v. and s.c.

SUMMARY:
The purpose of this study was to generate 16-week efficacy data, as well as up to 3-year efficacy, safety and tolerability data in subjects with active AS despite current or previous NSAID, DMARD and/or anti-TNF therapy.

ELIGIBILITY:
Inclusion criteria: moderate to severe AS, prior radiographic evidence according to the Modified NY Criteria (1984), inadequate response to NSAIDs. -- Exclusion criteria: pregnancy or lactation, on-going infectious or malignant process on a chest X-ray or MRI, previous exposure to IL-17 or IL-17R targeting therapies, previous exposure to any biological immunomodulating agent excluding TNF antagonists, previous cell depleting therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2015-02-23 (Actual); Study Completion 2017-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (51):
- United States (14):
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Peoria, Arizona
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Palm Harbor, Florida
  - Novartis Investigative Site, Pembroke Pines, Florida
  - Novartis Investigative Site, Passaic, New Jersey
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Mesquite, Texas
- Belgium (2):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brussels
- Czechia (2):
  - Novartis Investigative Site, Uherské Hradiště, Czech Republic
  - Novartis Investigative Site, Prague
- Germany (12):
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Zerbst
- Greece (4):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Heraklion
- Mexico (3):
  - Novartis Investigative Site, Torreón, Coahuila
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Culiacan, State of Mexico
- Portugal (2):
  - Novartis Investigative Site, Almada
  - Novartis Investigative Site, Lisbon
- Russia (3):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (6):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Madrid
- United Kingdom (3):
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Torquay

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] Dougados M, Kiltz U, Kivitz A, Pavelka K, Rohrer S, McCreddin S, Quebe-Fehling E, Porter B, Talloczy Z. Nonsteroidal anti-inflammatory drug-sparing effect of secukinumab in patients with radiographic axial spondyloarthritis: 4-year results from the MEASURE 2, 3 and 4 phase III trials. Rheumatol Int. 2022 Feb;42(2):205-213. doi: 10.1007/s00296-021-05044-6. Epub 2021 Nov 13. PMID 34773130
- [Derived] van der Horst-Bruinsma I, Miceli-Richard C, Braun J, Marzo-Ortega H, Pavelka K, Kivitz AJ, Deodhar A, Bao W, Porter B, Pournara E. A Pooled Analysis Reporting the Efficacy and Safety of Secukinumab in Male and Female Patients with Ankylosing Spondylitis. Rheumatol Ther. 2021 Dec;8(4):1775-1787. doi: 10.1007/s40744-021-00380-2. Epub 2021 Oct 7. PMID 34618347
- [Derived] Schett G, Baraliakos X, Van den Bosch F, Deodhar A, Ostergaard M, Gupta AD, Mpofu S, Fox T, Winseck A, Porter B, Shete A, Gensler LS. Secukinumab Efficacy on Enthesitis in Patients With Ankylosing Spondylitis: Pooled Analysis of Four Pivotal Phase III Studies. J Rheumatol. 2021 Aug;48(8):1251-1258. doi: 10.3899/jrheum.201111. Epub 2021 Mar 15. PMID 33722947
- [Derived] Deodhar AA, Miceli-Richard C, Baraliakos X, Marzo-Ortega H, Gladman DD, Blanco R, Das Gupta A, Martin R, Safi J Jr, Porter B, Shete A, Rosenbaum JT. Incidence of Uveitis in Secukinumab-treated Patients With Ankylosing Spondylitis: Pooled Data Analysis From Three Phase 3 Studies. ACR Open Rheumatol. 2020 May;2(5):294-299. doi: 10.1002/acr2.11139. Epub 2020 Apr 30. PMID 32352653
- [Derived] Deodhar A, Gladman DD, McInnes IB, Spindeldreher S, Martin R, Pricop L, Porter B, Safi J Jr, Shete A, Bruin G. Secukinumab Immunogenicity over 52 Weeks in Patients with Psoriatic Arthritis and Ankylosing Spondylitis. J Rheumatol. 2020 Apr;47(4):539-547. doi: 10.3899/jrheum.190116. Epub 2019 Jun 15. PMID 31203228
- [Derived] Pavelka K, Kivitz A, Dokoupilova E, Blanco R, Maradiaga M, Tahir H, Pricop L, Andersson M, Readie A, Porter B. Efficacy, safety, and tolerability of secukinumab in patients with active ankylosing spondylitis: a randomized, double-blind phase 3 study, MEASURE 3. Arthritis Res Ther. 2017 Dec 22;19(1):285. doi: 10.1186/s13075-017-1490-y. PMID 29273067
- See also: Introduction to clinical trials conducted by Novartis and to results of completed studies, with the aim of increasing the transparency of Novartis clinical research and making publicly available objective scientific information in a standardised format. — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to one of three treatment groups (1:1:1) and planned to be treated for 156 weeks. At Week 16, subjects who were randomized to placebo were re-randomized to secukinumab 150 mg or 300 mg. Patients were enrolled in 54 centers in Germany, Spain, United States, Czech Republic, Belgium, Greece, Mexico, Portugal, Russia and UK.
Pre-assignment Details: A screening period (SCR) running up to 10 weeks before randomization was used to assess eligibility.
Groups:
- Placebo i.v. and s.c.: Three i.v. infusions: at Baseline and weeks 2 and 4, followed by one s.c. injection at weeks 8 and 12. At week 16, 36 patients were re-randomised to Secukinumab 150mg and 37 patients to Secukinumab 300mg until the end of the study.
Period: Primary Assessment (up to Week 16)
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Started (Randomized set comprised all randomized patients) | 74 | 76 | 76
FAS (Full Analysis Set (FAS) all patients randomized and study treatment assigned.) | 74 | 76 | 76
Safety Set (all patients who received at least one dose of study treatment) | 74 | 76 | 75
Completed | 74 | 75 | 73
Not Completed | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 3
Period: Week 16 - 156
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Started | 74 | 75 | 73
Completed | 55 | 62 | 63
Not Completed | 19 | 13 | 10
Not completed — Adverse Event | 4 | 2 | 3
Not completed — Withdrawal by Subject | 7 | 3 | 5
Not completed — No longer requires treatment | 0 | 1 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Lack of Efficacy | 3 | 5 | 2
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c. | Total
Number analyzed (Participants) | 74 | 76 | 76 | 226
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.9 (11.11) | 42.1 (11.81) | 42.7 (11.43) | 42.5 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 36 | 90
  Male | 46 | 50 | 40 | 136
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 54 | 52 | 58 | 164
  Black or African American | 2 | 2 | 1 | 5
  Asian | 1 | 2 | 0 | 3
  American Indian or Alaska Native | 4 | 6 | 5 | 15
  Unknown | 0 | 1 | 0 | 1
  Other | 13 | 13 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 20% Improvement in the Assessment of Spondyloarthritis International Society Criteria Scale / ASAS 20 Response
Description: ASAS 20 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame at least 20% improvement in score in at least 3 of a conventional set of 4 clinical domains relevant to AS and no worsening in the fourth domain. In this study, ASAS 20 was used to assess the efficacy of at least one dose of secukinumab versus placebo.
Time Frame: 16 weeks
Population: FAS - Missing ASAS responses were considered as non-responder
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Number analyzed (Participants) | 74 | 76 | 76
Participants
  Responder | 43 | 46 | 28
  Non-Responder | 31 | 30 | 48
Statistical Analysis 1: Comparison: Secukinumab 10 mg/kg i.v. / 150 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0093, Regression, Logistic; Odds Ratio (OR) = 2.41, 95% CI 2-sided [1.24 to 4.69]
Statistical Analysis 2: Comparison: Secukinumab 10 mg/kg i.v. / 300 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0037, Regression, Logistic; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.38 to 5.21]

2. Secondary Outcome: ASAS 40 Response
Description: ASAS 40 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame at least 40% improvement in score in at least 3 of a conventional set of 4 clinical domains relevant to AS and no worsening in the fourth domain. In this study, ASAS 40 was used to assess the efficacy of at least one dose of secukinumab versus placebo.
Time Frame: 16 weeks
Population: FAS - Missing ASAS responses were considered as non-responder
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Number analyzed (Participants) | 74 | 76 | 76
Participants
  Responder | 30 | 32 | 16
  Non-Responder | 44 | 44 | 60
Statistical Analysis 1: Comparison: Secukinumab 10 mg/kg i.v. / 150 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0100, Regression, Logistic; Odds Ratio (OR) = 2.59, 95% CI 2-sided [1.26 to 5.35]
Statistical Analysis 2: Comparison: Secukinumab 10 mg/kg i.v. / 300 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0051, Regression, Logistic; Odds Ratio (OR) = 2.81, 95% CI 2-sided [1.36 to 5.78]

3. Secondary Outcome: Serum hsCRP
Description: Blood levels of C-reactive protein (CRP), an acute phase reactant, are indicative of inflammation and of its severity, and can be used to monitor treatment response. A high sensitivity CRP (hsCRP) test was implemented in this study, to assess the efficacy of at least one dose of secukinumab versus placebo in reducing AS elicited systemic inflammation over the time.
Time Frame: Baseline and 16 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Number analyzed (Participants) | 74 | 76 | 76
mg/L
  Baseline | 15.79 (21.075) | 11.08 (13.285) | 13.91 (19.999)
  Week 16: number analyzed (Participants) | 72 | 74 | 70
  Week 16 | 7.68 (13.277) | 4.34 (5.433) | 15.34 (21.694)
  Change from Baseline to Week 16 | -8.06 (21.132) | -6.75 (13.778) | 0.57 (11.629)
Statistical Analysis 1: Comparison: Secukinumab 10 mg/kg i.v. / 150 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Relative treatment effect = 0.51, 95% CI 2-sided [0.38 to 0.68] — Relative treatment effect = exponential of the difference in LSM on the log e scale or the geometric LSM ratio on the original scale. For values less than 1, AIN457 has a greater reduction than Placebo
Statistical Analysis 2: Comparison: Secukinumab 10 mg/kg i.v. / 300 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Relative treatment effect = 0.44, 95% CI 2-sided [0.33 to 0.60] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: ASAS 5/6 Response
Description: ASAS 5/6 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame at least 20% improvement in score in at least 5 of a conventional set of 6 clinical domains relevant to AS and no worsening in the remaining domain. In this study, ASAS 5/6 was used to assess the efficacy of at least one dose of secukinumab versus placebo.
Time Frame: 16 weeks
Population: FAS - Missing ASAS responses were considered as non-responder
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Number analyzed (Participants) | 74 | 76 | 76
Participants
  Responder | 31 | 30 | 11
  Non-Responder | 43 | 46 | 65
Statistical Analysis 1: Comparison: Secukinumab 10 mg/kg i.v. / 150 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 4.46, 95% CI 2-sided [2.01 to 9.92]
Statistical Analysis 2: Comparison: Secukinumab 10 mg/kg i.v. / 300 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 4.21, 95% CI 2-sided [1.89 to 9.38]

5. Secondary Outcome: Bath Ankylosing Spondylitis Disease Activity Index / BASDAI
Description: BASDAI is a validated assessment tool using 0 through 10 scales (0 indicating "no problem" and 10 indicating "worst problem"), to characterise six clinical domains pertaining to five major symptoms of AS perceived by the patients. Computed composite scores of 4 or greater indicate suboptimal disease control. In this study, the BASDAI index was used to assess the efficacy of at least one dose of secukinumab versus placebo.
Time Frame: Baseline and 16 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Number analyzed (Participants) | 74 | 76 | 76
units on a scale
  Baseline | 6.958 (1.3913) | 6.963 (1.3766) | 6.907 (1.2600)
  Week 16: number analyzed (Participants) | 72 | 73 | 70
  Week 16 | 4.451 (2.5623) | 4.178 (2.7038) | 5.369 (2.2574)
  Change from Baseline to Week 16: number analyzed (Participants) | 72 | 73 | 70
  Change from Baseline to Week 16 | -2.548 (2.4559) | -2.796 (2.6374) | -1.590 (2.0084)
Statistical Analysis 1: Comparison: Secukinumab 10 mg/kg i.v. / 150 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0347, Mixed Models Analysis; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.60 to -0.06], Standard Error of Mean 0.390
Statistical Analysis 2: Comparison: Secukinumab 10 mg/kg i.v. / 300 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0018, Mixed Models Analysis; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-2.00 to -0.46], Standard Error of Mean 0.390

6. Secondary Outcome: Number of Participants With Successful Self-administration (to Measure Usability of Pre-filled Syringe)
Description: Successful self-administration is defined as success in steps P8 (Removed Needle Cap from Safety Syringe), P10 (Pinched the Skin at Injection Site), P11 (Inserted the Needle into Skin), P12 (Held onto the Finger Flange), P13 (Fully Depressed Plunger until End Point), and P14 (Held Plunger Down and Syringe in Place) of the Instructions for Use, as observed by the site staff at applicable visits.
Time Frame: Week 8 and Week 12
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Number analyzed (Participants) | 74 | 76 | 75
Participants
  Self-administration Week 8: Successful Self-administration | 72 | 73 | 71
  Self-administration Week 8: Unsuccessful Self-administration | 0 | 0 | 1
  Self-administration Week 8: Missing | 2 | 3 | 3
  Self-administration Week 12: Successful Self-administration | 74 | 75 | 72
  Self-administration Week 12: Unsuccessful Self-administration | 0 | 0 | 0
  Self-administration Week 12: Missing | 0 | 1 | 3

7. Secondary Outcome: Pre-filled Syringe Possible Hazard
Description: The number and percentage of subjects who experience any of the defined possible hazards are summarized, as defined in the Possible Hazard assessment check list and as observed by the site staff at applicable visits.
Time Frame: Week 8 and Week 12
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Number analyzed (Participants) | 74 | 76 | 75
Participants
  Week 8:Was needle stick in a critical area?: Yes | 0 | 0 | 0
  Week 8:Was needle stick in a critical area?: No | 73 | 73 | 72
  Week 8:Was needle stick in a critical area?: Missing | 1 | 3 | 3
  Week 8: Was needle stick in a non-critical area?: Yes | 2 | 5 | 3
  Week 8: Was needle stick in a non-critical area?: No | 71 | 68 | 69
  Week 8: Was needle stick in a non-critical area?: Missing | 1 | 3 | 3
  Week 8: Was any part of the device swallowed?: Yes | 0 | 0 | 0
  Week 8: Was any part of the device swallowed?: No | 73 | 73 | 72
  Week 8: Was any part of the device swallowed?: Missing | 1 | 3 | 3
  Week 8: Was allergic reaction to device noticed?: Yes | 0 | 0 | 0
  Week 8: Was allergic reaction to device noticed?: No | 73 | 73 | 72
  Week 8: Was allergic reaction to device noticed?: Missing | 1 | 3 | 3
  Week 8: Was pain increased due to bent needle?: Yes | 0 | 0 | 0
  Week 8: Was pain increased due to bent needle?: No | 73 | 73 | 72
  Week 8: Was pain increased due to bent needle?: Missing | 1 | 3 | 3
  Week 8: Was there breakage of device observed?: Yes | 0 | 0 | 0
  Week 8: Was there breakage of device observed?: No | 73 | 73 | 72
  Week 8: Was there breakage of device observed?: Missing | 1 | 3 | 3
  Week 8:Was swallowing of debris observed?: Yes | 0 | 0 | 0
  Week 8:Was swallowing of debris observed?: No | 73 | 73 | 72
  Week 8:Was swallowing of debris observed?: Missing | 1 | 3 | 3
  Week 8:Was any other problem observed?: Yes | 1 | 0 | 0
  Week 8:Was any other problem observed?: No | 72 | 73 | 72
  Week 8:Was any other problem observed?: Missing | 1 | 3 | 3
  Week 8:Was less than the full dose administered: Yes | 0 | 0 | 0
  Week 8:Was less than the full dose administered: No | 73 | 73 | 72
  Week 8:Was less than the full dose administered: Missing | 1 | 3 | 3
  Week 12: Was needle stick in a critical area?: Yes | 0 | 0 | 0
  Week 12: Was needle stick in a critical area?: No | 74 | 75 | 72
  Week 12: Was needle stick in a critical area?: Missing | 0 | 1 | 3
  Week 12: Was needle stick in a non-critical area?: Yes | 1 | 4 | 3
  Week 12: Was needle stick in a non-critical area?: No | 73 | 71 | 69
  Week 12: Was needle stick in a non-critical area?: Missing | 0 | 1 | 3
  Week 12: Was any part of the device swallowed?: Yes | 0 | 0 | 0
  Week 12: Was any part of the device swallowed?: No | 74 | 75 | 72
  Week 12: Was any part of the device swallowed?: Missing | 0 | 1 | 3
  Week 12: Was allergic reaction to device noticed?: Yes | 0 | 0 | 0
  Week 12: Was allergic reaction to device noticed?: No | 74 | 75 | 72
  Week 12: Was allergic reaction to device noticed?: Missing | 0 | 1 | 3
  Week 12: Was pain increased due to bent needle?: Yes | 0 | 0 | 0
  Week 12: Was pain increased due to bent needle?: No | 74 | 75 | 72
  Week 12: Was pain increased due to bent needle?: Missing | 0 | 1 | 3
  Week 12: Was there breakage of device observed?: Yes | 0 | 0 | 0
  Week 12: Was there breakage of device observed?: No | 74 | 75 | 72
  Week 12: Was there breakage of device observed?: Missing | 0 | 1 | 3
  Week 12: Was swallowing of debris observed?: Yes | 0 | 0 | 0
  Week 12: Was swallowing of debris observed?: No | 74 | 75 | 72
  Week 12: Was swallowing of debris observed?: Missing | 0 | 1 | 3
  Week 12: Was any other problem observed?: Yes | 1 | 1 | 0
  Week 12: Was any other problem observed?: No | 73 | 74 | 72
  Week 12: Was any other problem observed?: Missing | 0 | 1 | 3
  Week 12: Was less than the full dose administered?: Yes | 0 | 0 | 0
  Week 12: Was less than the full dose administered?: No | 74 | 75 | 72
  Week 12: Was less than the full dose administered?: Missing | 0 | 1 | 3

8. Secondary Outcome: Prefilled Syringe Patient Satisfaction Assessment
Description: The self-injection assessment questionnaire (SIAQ) measures overall patient experience with subcutaneous self-injection at applicable visits. Domain scores ranging from 0 (worst experience) to 10 (best experience) are presented: Feeling about injections, Self-confidence, Satisfaction with self-injection.
Time Frame: Baseline, weeks 8, 12 and 16
Population: Safety Set
Measure: Mean (Standard Deviation); unit: Points
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Number analyzed (Participants) | 74 | 76 | 75
Points
  Week 0: Feeling about injections | 7.97 (1.946) | 7.66 (2.369) | 8.01 (1.927)
  Week 8: Feeling about injections: number analyzed (Participants) | 73 | 73 | 71
  Week 8: Feeling about injections | 7.96 (2.538) | 7.68 (2.296) | 8.24 (2.082)
  Week 12: Feeling about injections: number analyzed (Participants) | 71 | 73 | 70
  Week 12: Feeling about injections | 8.45 (1.968) | 7.93 (2.201) | 8.25 (1.997)
  Week 16: Feeling about injections: number analyzed (Participants) | 71 | 71 | 73
  Week 16: Feeling about injections | 8.15 (2.337) | 7.99 (2.269) | 8.41 (2.037)
  Week 0: Self-confidence | 6.27 (2.811) | 6.66 (2.315) | 6.52 (2.273)
  Week 8: Self-confidence: number analyzed (Participants) | 73 | 73 | 71
  Week 8: Self-confidence | 7.08 (2.520) | 6.66 (2.855) | 7.41 (2.198)
  Week 12: Self-confidence: number analyzed (Participants) | 71 | 73 | 70
  Week 12: Self-confidence | 7.01 (2.603) | 7.28 (2.231) | 7.42 (2.230)
  Week 16: Self-confidence: number analyzed (Participants) | 71 | 71 | 73
  Week 16: Self-confidence | 7.51 (2.388) | 7.23 (2.566) | 7.64 (2.192)
  Week 0: Satisfaction with self-injection | 5.34 (2.692) | 6.12 (2.429) | 5.30 (2.694)
  Week 8: Satisfaction with self-injection: number analyzed (Participants) | 73 | 73 | 71
  Week 8: Satisfaction with self-injection | 7.67 (1.734) | 7.50 (1.667) | 7.39 (2.002)
  Week 12: Satisfaction with self-injection: number analyzed (Participants) | 71 | 73 | 70
  Week 12: Satisfaction with self-injection | 7.68 (1.483) | 7.50 (1.816) | 7.46 (1.780)
  Week 16: Satisfaction with self-injection: number analyzed (Participants) | 71 | 71 | 73
  Week 16: Satisfaction with self-injection | 7.57 (1.741) | 7.82 (1.933) | 7.67 (1.577)

9. Secondary Outcome: ASAS Partial Remission
Description: ASAS partial remission is a composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame a value not above 2 units in each of the 4 ASAS domains on a scale of 10. In this study, ASAS partial remission was used to assess the efficacy of at least one dose of secukinumab versus placebo.
Time Frame: 16 weeks
Population: FAS - Missing ASAS responses were considered as non-responder
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 10 mg/kg i.v. / 150 mg s.c. | Secukinumab 10 mg/kg i.v. / 300 mg s.c. | Placebo i.v. and s.c.
Number analyzed (Participants) | 74 | 76 | 76
Participants
  Responder | 7 | 16 | 1
  Non-Responder | 67 | 60 | 75
Statistical Analysis 1: Comparison: Secukinumab 10 mg/kg i.v. / 150 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0593, Regression, Logistic; Odds Ratio (OR) = 7.71, 95% CI 2-sided [0.92 to 64.42]
Statistical Analysis 2: Comparison: Secukinumab 10 mg/kg i.v. / 300 mg s.c. vs Placebo i.v. and s.c; Test type: Superiority; p = 0.0046, Regression, Logistic; Odds Ratio (OR) = 19.39, 95% CI 2-sided [2.49 to 150.79]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 3 years.
Description: Patients randomized to Placebo at Baseline are reported under Placebo for AEs starting before re-randomization to Secukinumab (Week 16) and under the respective Secukinumab arm for AEs starting after re-randomization to Secukinumab (Week 16).
Groups:
- Any Secukinumab 150 mg: Includes Patients randomized to Secukinumab 150 mg at baseline + patients re-randomized to Secukinumab 150 mg at week 16 (for AEs occurring after rerandomization)
- Any Secukinumab 300 mg: Includes Patients randomized to Secukinumab 300 mg at baseline + patients re-randomized to Secukinumab 300 mg at week 16 (for AEs occurring after rerandomization)
- Any Secukinumab: Any Secukinumab 150 mg + Any Secukinumab 300 mg
- Placebo: Includes Patients randomized to Placebo for AEs until time of re-randomization (Week 16) to Secukinumab.
Arm/Group | Any Secukinumab 150 mg | Any Secukinumab 300 mg | Any Secukinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/113 | 0/223 | 0/75
Serious Adverse Events (participants affected / at risk) | 11/110 | 11/113 | 22/223 | 1/75
Other Adverse Events (participants affected / at risk) | 86/110 | 89/113 | 175/223 | 28/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any Secukinumab 150 mg (N=110) | Any Secukinumab 300 mg (N=113) | Any Secukinumab (N=223) | Placebo (N=75)
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 1 | 1 | 0
Vogt-Koyanagi-Harada syndrome (Eye disorders) | 0 | 1 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 1 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any Secukinumab 150 mg (N=110) | Any Secukinumab 300 mg (N=113) | Any Secukinumab (N=223) | Placebo (N=75)
Iritis (Eye disorders) | 0 | 3 | 3 | 0
Uveitis (Eye disorders) | 3 | 5 | 8 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 11 | 9 | 20 | 0
Food poisoning (Gastrointestinal disorders) | 2 | 3 | 5 | 0
Gastritis (Gastrointestinal disorders) | 3 | 1 | 4 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 7 | 1
Toothache (Gastrointestinal disorders) | 3 | 2 | 5 | 1
Vomiting (Gastrointestinal disorders) | 0 | 4 | 4 | 0
Fatigue (General disorders) | 5 | 4 | 9 | 0
Influenza like illness (General disorders) | 2 | 1 | 3 | 2
Bronchitis (Infections and infestations) | 14 | 9 | 23 | 1
Conjunctivitis (Infections and infestations) | 1 | 3 | 4 | 1
Ear infection (Infections and infestations) | 0 | 3 | 3 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 3 | 4 | 0
Influenza (Infections and infestations) | 3 | 9 | 12 | 0
Nasopharyngitis (Infections and infestations) | 27 | 27 | 54 | 2
Oral herpes (Infections and infestations) | 1 | 3 | 4 | 1
Pharyngitis (Infections and infestations) | 3 | 6 | 9 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 3 | 3 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 4 | 0
Pulpitis dental (Infections and infestations) | 4 | 1 | 5 | 2
Respiratory tract infection (Infections and infestations) | 12 | 10 | 22 | 4
Rhinitis (Infections and infestations) | 6 | 4 | 10 | 0
Sinusitis (Infections and infestations) | 8 | 1 | 9 | 2
Tonsillitis (Infections and infestations) | 4 | 4 | 8 | 0
Upper respiratory tract infection (Infections and infestations) | 12 | 16 | 28 | 2
Urinary tract infection (Infections and infestations) | 4 | 6 | 10 | 2
Sunburn (Injury, poisoning and procedural complications) | 0 | 3 | 3 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 5 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 3 | 7 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 13 | 27 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 3 | 7 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 12 | 19 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5 | 8 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4 | 0
Dizziness (Nervous system disorders) | 2 | 4 | 6 | 1
Headache (Nervous system disorders) | 12 | 14 | 26 | 5
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 2 | 2
Migraine (Nervous system disorders) | 5 | 1 | 6 | 0
Paraesthesia (Nervous system disorders) | 4 | 0 | 4 | 0
Depression (Psychiatric disorders) | 3 | 3 | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 12 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 14 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 4 | 0
Hypertension (Vascular disorders) | 7 | 5 | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.